CLINICAL TRIAL: NCT00280280
Title: Double-blind Comparison of Botox Versus Baclofen for the Treatment of Subjects With Upper Limb Spasticity - Pilot Study
Brief Title: Botox vs. Baclofen for Upper Limb Spasticity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low patient accrual
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, David Charles, Associate Professor Neurology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 050935
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Spasticity
Keywords: spasticity; Botox; baclofen
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): This study will explore the safety and effectiveness of Botox versus baclofen in treatment subjects with upper-limb spasticity due to neurological damage or a stable neurological disorder. Subjects will be randomized to one of two treatment groups: intramuscular Botox plus oral placebo or intramuscular placebo plus oral baclofen.
  Interventions: Drug: intramuscular Botox versus oral baclofen

INTERVENTIONS:
Drug: intramuscular Botox versus oral baclofen — Each vial of Botox contains 100 units of Clostridium botulinum toxin type A, 0.5 mg albumin (human) and 0.9 mg sodium chloride in a sterile, vacuum-dried form without a preservative. Botox placebo is sterile normal saline (without preservatives) for injection. Baclofen is supplied as 10 mg tablets for oral administration. Inactive ingredients include colloidal anhydrous silica, microcrystalline cellulose, magnesium stearate, povidone, wheat starch. Baclofen placebo tablets are composed of microcrystalline cellulose binder (99%), magnesium stearate 0.5%, and silica gel 0.5% and appear similar to commercial Baclofen tablets.

SUMMARY:
The purposes of this pilot study are to evaluate the safety and efficacy of Botox® compared to the safety and efficacy of oral baclofen in reducing muscle tone-related disability resulting from neurological damage or a stable neurological disorder and to evaluate drug-therapy tolerance.

DETAILED DESCRIPTION:
Spasticity results from any injury to the central nervous system, including brain or spinal cord. Illnesses or injuries that typically cause spasticity include cerebral palsy, stroke, multiple sclerosis and traumatic brain or spinal cord injury. Common treatments for spasticity include physical and occupational therapy as well as oral medications such as baclofen, injected medications such as botulinum neurotoxin, intrathecal medications and surgical procedures. The approach to the treatment of spasticity is comprehensive in nature and these therapies have been widely applied to a broad population of patients including children, adults and older adults.

This is a single-center, randomized, prospective, parallel, double-blind study. Study duration is approximately 16 weeks.At Visit 2 (Baseline Visit), all eligible study subjects will be randomized to one of two treatment groups: intramuscular Botox plus oral placebo, or intramuscular placebo plus oral baclofen.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female subjects of any race, and at least 18 years of age. Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline (test must have a sensitivity of at least 50mlU/ml for human chorionic gonadotropin) and practice a reliable method of contraception throughout the study;
* Minimal 4-month history stable neurological disorder resulting focal upper limb muscle spasticity (wrist and/or elbow)
* Disability Assessment Scale (DAS) ≥ 2 for the principal therapeutic intervention target as chosen by Investigator and Subject (i.e., hygiene, dressing, pain and cosmesis).
* Subjects who are able to understand the requirements of the study and sign Informed Consent/HIPAA Authorization forms.

Exclusion Criteria:

* Female subjects who are pregnant (positive urine pregnancy test) or who have an infant they are breast-feeding or who are of childbearing potential and are not practicing a reliable method of birth control.
* Severe contracture at the wrist or a history of tendon transfer in the study limb.
* Cast of study limb within four weeks of Visit 1.
* Profound atrophy of the muscles in the target area(s) of injection.
* Progressive neurological disorder (e.g., multiple sclerosis).
* Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis or any other disease that might interfere with neuromuscular function.
* Orthostatic hypotension or current use of alpha-2 adrenergic agonists (e.g. clonidine).
* Current anticoagulant therapy and INR > 3.5
* Significantly impaired renal and/or hepatic function, in the opinion of the Investigator.
* Failure to meet prohibited concomitant medication criteria (Supplement I)
* Subjects planning inpatient surgery during the study.
* Any uncontrolled systemic disease.
* Allergy or sensitivity to any component of the study medication.
* Recent alcohol or drug abuse.
* History of poor cooperation, non-compliance with medical treatment, or unreliability.
* Subjects currently participating in an investigational drug study or who have participated in an investigational drug study within 30 days of the Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Disability Assessment Scale (DAS) | 4 months

SECONDARY OUTCOMES:
Modified Ashworth Tone | 4 months
Subject Questionnaires | 4 months
Contralateral Finger Tap Test | 4 months
Contralateral Grip Strength | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: P. David Charles, MD, Principal Investigator — Vanderbilt University Department of Neurology
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States